CLINICAL TRIAL: NCT03453658
Title: Evaluation of Mechanized Instrumentation for Endodontic Treatment of Primary Teeth - Randomized Clinical Trial
Brief Title: Mechanized Instrumentation for Endodontic Treatment of Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fausto Medeiros Mendes, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FOUSP2912
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Endodontic Treatment of Primary Teeth
Keywords: Endodontics; Primary Teeth; Reciprocating instrumentation; Mechanized instrumentation

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, controlled clinical trial with two parallel arms.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be a different examiner who will be unaware of the allocated group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual instrumentation (Active Comparator): Manual instrumentation: Endodontic treatment will be performed with the use of conventional endodontic manual files.
  Interventions: Procedure: Manual instrumentation
- Reciprocating instrumentation (Experimental): Mechanized instrumentation: Endodontic treatment will be performed with the use of reciprocating mechanized files. The files are activated by an engine that produces reciprocating movements.
  Interventions: Procedure: Reciprocating Instrumentation

INTERVENTIONS:
Procedure: Manual instrumentation — Manual conventional files will be used in endodontic treatment of primary teeth
  Arms: Manual instrumentation
Procedure: Reciprocating Instrumentation — Reciprocating files system will be used in endodontic treatment of primary teeth.
  Arms: Reciprocating instrumentation

SUMMARY:
Mechanized instrumentation systems stand out amongst various devices used in modern Endodontics. Its use in Pediatric Dentistry, its action in primary teeth, has been in the center of many discussions and laboratory studies. Nevertheless, up to now, a lack of clinical studies on this issue can be found. Our objective is to conduct a double blinded, 2 years follow up clinical trial to compare the success of endodontic treatment in primary teeth using mechanized reciprocating instrumentation to the use of manual instrumentation.

DETAILED DESCRIPTION:
With the approval of the Ethics Committee of University of São Paulo, after clinical and radiographic examination, patients in search for endodontic treatment in primary teeth will be invited to take part in the study. The participants of the study will be randomized to one of two groups (manual or reciprocating instrumentation). Endodontic treatment will be held by a specialist according to the randomized group. A blinded examiner will proceed one week, 3 months, 6 months, 12 months and 24 months follow ups. Clinical and radiographic conditions of endodontic treatments will be analyzed to classify them as Success or Failure. The unit of analysis will be the teeth; hence, each participant may have more than one tooth included in the study. The randomization will be performed considering the tooth. Data analysis will consider the cluster nature of the sample.

The primary outcome of the study will be the success rates according to the groups. The longevity of treatments will be evaluated by estimating survival rates by Kaplan-Meier and Cox regression. The differences between survival rates of both groups will be through Cox regression adjusted for the cluster nature of the sample (more than one tooth per participant), considering a level of significance of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Primary molar teeth with necessity of endodontic treatment.
* Patients whose parents or guardians consent to their participation in the study

Exclusion Criteria:

Teeth presenting one of the following:

* Resorption of more than 2/3 of the root
* Destruction of the crypt of the permanent successor
* Pulp chamber floor drilling.
* Presence of internal resorption

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Success or failure of endodontic treatment | Two years
  The success or failure of endodontic treatments evaluated by the time spent in the tooth arch in clinical conditions of normality. Clinical criteria for determining success are: absence of fistula, absence of painful symptoms and pathological absence of adequate mobility and gingival contour. Radiographically, the success criteria are: absence / reduction of periapical bone rarefaction in anterior and absence / bone rarefaction in the furcation area of later, maintaining the periradicular space, root resorption compatible with the eruptive phase and absence of pathological bone resorption. To evaluate the reduction of lesions or appearance of new lesions will be between the initial and follow-up radiographs. Radiographs will be scanned and the end of the bone rarefactions starting area and will be measured on a software image analysis.

SECONDARY OUTCOMES:
Appointment duration | After treatment
  The time spent using both techniques will be measured and compared between the groups. The time will be recorded in minutes since the end of anesthesia and rubber-dam placement until the beginning of restorative procedure.
Quality of obturation provided by two different instrumentation techniques | After treatment
  After root canal obturation, a final periapical radiograph will be digitalized and analyzed, obtaining the percentage of root canal filling provided by each instrumentation technique.
Discomfort related to each instrumentation technique | After treatment.
  Discomfort provided by each technique will be analyzed and compared between the groups using a validated facial scale, named Wong-Baker facial scale. This is a scale of 6 drawn faces ranging from a smiling representing no hurt face to as crying hurts worst face. Therefore, the scale has been used to evaluate pain and/or discomfort after several procedures, including dental procedures. The answers can be measured as a qualitative ordinal variable varying from 0 (no hurt) to 5 (Hurts worst). This scale has been used previously in pediatric dentistry context (Tomlinson et al., 2010).
Cost-Efficacy of each instrumentation technique | Two years
  The cost-efficacy of each procedure will be analyzed according to the success rate of each technique, and the results obtained will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Renata Marques, PhD Student, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Dentistry, University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
We are planning to share the individual data upon request, since the participants and their legal guardians consent.

REFERENCES:
- [Background] Ahmad IA, Pani SC. Accuracy of electronic apex locators in primary teeth: a meta-analysis. Int Endod J. 2015 Mar;48(3):298-307. doi: 10.1111/iej.12315. Epub 2014 Jun 28. PMID 24863852
- [Background] Ahmed HM. Anatomical challenges, electronic working length determination and current developments in root canal preparation of primary molar teeth. Int Endod J. 2013 Nov;46(11):1011-22. doi: 10.1111/iej.12134. Epub 2013 May 25. PMID 23711096
- [Background] Canoglu H, Tekcicek MU, Cehreli ZC. Comparison of conventional, rotary, and ultrasonic preparation, different final irrigation regimens, and 2 sealers in primary molar root canal therapy. Pediatr Dent. 2006 Nov-Dec;28(6):518-23. PMID 17249433
- [Background] Fumes AC, Sousa-Neto MD, Leoni GB, Versiani MA, da Silva LA, da Silva RA, Consolaro A. Root canal morphology of primary molars: a micro-computed tomography study. Eur Arch Paediatr Dent. 2014 Oct;15(5):317-26. doi: 10.1007/s40368-014-0117-0. Epub 2014 Feb 22. PMID 24563173
- [Background] Kummer TR, Calvo MC, Cordeiro MM, de Sousa Vieira R, de Carvalho Rocha MJ. Ex vivo study of manual and rotary instrumentation techniques in human primary teeth. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2008 Apr;105(4):e84-92. doi: 10.1016/j.tripleo.2007.12.008. PMID 18329573
- [Background] Fuks AB. Pulp therapy for the primary and young permanent dentitions. Dent Clin North Am. 2000 Jul;44(3):571-96, vii. PMID 10925773
- [Background] Lee GH, McGrath C, Yiu CK. Developing clinical practice guidelines for caries prevention and management for pre-school children through the ADAPTE process and Delphi consensus. Health Res Policy Syst. 2016 Jun 14;14(1):44. doi: 10.1186/s12961-016-0117-0. PMID 27301382
- [Background] Moura-Netto C, Palo RM, Pinto LF, Mello-Moura AC, Daltoe G, Wilhelmsen NS. CT study of the performance of reciprocating and oscillatory motions in flattened root canal areas. Braz Oral Res. 2015;29:1-6. doi: 10.1590/1807-3107bor-2015.vol29.0006. Epub 2014 Dec 2. PMID 25466329
- [Background] Nagaratna PJ, Shashikiran ND, Subbareddy VV. In vitro comparison of NiTi rotary instruments and stainless steel hand instruments in root canal preparations of primary and permanent molar. J Indian Soc Pedod Prev Dent. 2006 Dec;24(4):186-91. doi: 10.4103/0970-4388.28075. PMID 17183182
- [Background] Neena IE, Ananthraj A, Praveen P, Karthik V, Rani P. Comparison of digital radiography and apex locator with the conventional method in root length determination of primary teeth. J Indian Soc Pedod Prev Dent. 2011 Oct-Dec;29(4):300-4. doi: 10.4103/0970-4388.86371. PMID 22016313
- [Background] Nobrega DF, Fernandez CE, Del Bel Cury AA, Tenuta LM, Cury JA. Frequency of Fluoride Dentifrice Use and Caries Lesions Inhibition and Repair. Caries Res. 2016;50(2):133-40. doi: 10.1159/000444223. Epub 2016 Mar 19. PMID 26992247
- [Background] Pinheiro SL, Araujo G, Bincelli I, Cunha R, Bueno C. Evaluation of cleaning capacity and instrumentation time of manual, hybrid and rotary instrumentation techniques in primary molars. Int Endod J. 2012 Apr;45(4):379-85. doi: 10.1111/j.1365-2591.2011.01987.x. Epub 2011 Dec 22. PMID 22188162
- [Background] Piovesan C, Mendes FM, Ferreira FV, Guedes RS, Ardenghi TM. Socioeconomic inequalities in the distribution of dental caries in Brazilian preschool children. J Public Health Dent. 2010 Fall;70(4):319-26. doi: 10.1111/j.1752-7325.2010.00191.x. PMID 20735719
- [Background] Prabhakar AR, Yavagal C, Dixit K, Naik SV. Reciprocating vs Rotary Instrumentation in Pediatric Endodontics: Cone Beam Computed Tomographic Analysis of Deciduous Root Canals using Two Single-file Systems. Int J Clin Pediatr Dent. 2016 Jan-Mar;9(1):45-9. doi: 10.5005/jp-journals-10005-1332. Epub 2016 Apr 22. PMID 27274155
- [Background] Rasquin LC, de Carvalho FB, Lima RK. In vitro evaluation of root canal preparation using oscillatory and rotary systems in flattened root canals. J Appl Oral Sci. 2007 Feb;15(1):65-9. doi: 10.1590/s1678-77572007000100014. PMID 19089103
- [Background] George S, Anandaraj S, Issac JS, John SA, Harris A. Rotary endodontics in primary teeth - A review. Saudi Dent J. 2016 Jan;28(1):12-7. doi: 10.1016/j.sdentj.2015.08.004. Epub 2015 Nov 22. PMID 26792964
- [Background] Srinivasan V, Patchett CL, Waterhouse PJ. Is there life after Buckley's Formocresol? Part I -- a narrative review of alternative interventions and materials. Int J Paediatr Dent. 2006 Mar;16(2):117-27. doi: 10.1111/j.1365-263X.2006.00688.x. PMID 16430526
- [Background] Waterhouse PJ, Nunn JH, Whitworth JM, Soames JV. Primary molar pulp therapy--histological evaluation of failure. Int J Paediatr Dent. 2000 Dec;10(4):313-21. doi: 10.1046/j.1365-263x.2000.00211.x. PMID 11310245
- [Background] Tomlinson D, von Baeyer CL, Stinson JN, Sung L. A systematic review of faces scales for the self-report of pain intensity in children. Pediatrics. 2010 Nov;126(5):e1168-98. doi: 10.1542/peds.2010-1609. Epub 2010 Oct 4. PMID 20921070